CLINICAL TRIAL: NCT05228080
Title: Predictive Study of Serum Endocan for Hemorrhagic Transformation After Reperfusion Therapies in Acute Ischemic Stroke
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KY20212167
Record Dates: First submitted 2021-11-14; First posted 2022-02-08 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2021-11

CONDITIONS: Acute Ischemic Stroke
Keywords: endocan; stroke; reperfusion; hemorrhage
MeSH Terms: conditions — Ischemic Stroke; Stroke; Hemorrhage

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- acute ischemic stroke
  Interventions: Diagnostic Test: enzyme-linked immunosorbent assay(ELISA)

INTERVENTIONS:
Diagnostic Test: enzyme-linked immunosorbent assay(ELISA) — Peripheral blood samples will be drawn from each patient at study entry (before reperfusion therapy) and at 12,24 hours after reperfusion therapy.Serum will be immediately separated by centrifugation at 3000 rpm for 15 minutes and stored at -80°C. Endocan,ICAM-1,VCAM-1,MMP-9 levels will be determined in duplicate by commercially available enzyme-linked immunosorbent assay (ELISA).

SUMMARY:
Stroke is the second largest cause of death globally after ischemic heart disease.Of the total number of prevalent strokes, 84.4% are ischemic. Reperfusion therapy is the most important treatment for acute ischemic stroke (AIS) ,including intravenous thrombolysis and/or endovascular treatment.However,the most serious and common complication with reperfusion therapy is hemorrhage transformation(HT),which significantly increases disability and mortality. The fundamental mechanism leading to post-stroke HT is the disruption of the blood brain barrier(BBB) and increase of permeability.Endocan plays a critical role in vascular inflammatory responses by enhances the production of pro-inflammatory cytokines by endothelial cells,the expression of adhesion molecules such as inter-cellular adhesion molecule-1(ICAM-1) and vascular cell adhesion molecule-1(VCAM-1),and the adhesion of leukocytes to endothelial cells. Endocan significantly decreases levels of zonula occludens（ZO-1) and occludin which are tight junction proteins that play major roles in the maintenance of vascular barriers. Endocan could induce vascular endothelial growth factor-A(VEGF-A) and facilitate the binding of VEGF-A to its receptor(VEGFR-2) to enhanced endothelial permeability.Therefore,endocan is a reliable biomarker of endothelial dysfunction, which may be associated with disruption of the BBB. In this context, the investigators hypothesized that elevated pretreatment serum endocan levels might be independently associated with HT after reperfusion therapy in the acute phase of ischemic stroke. Serum endocan,ICAM-1,VCAM-1 and matrix metalloproteinase-9(MMP-9) levels will be determined by enzyme-linked immunosorbent assay(ELISA) in blood samples obtained at baseline (pretreatment) and at 12,24 hours after reperfusion therapy in patients with acute stroke and in healthy subjects.In the present study,the investigators attempt to investigate whether high levels of endocan are associated with HT in patients who received reperfusion therapy.In addition,the investigators explore the association between serum endocan and early neurological deterioration and unfavourable short-term prognosis.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of acute ischemic stroke and presentation at the hospital within 24h from symptom onset
* Eligibility for intravenous thrombolysis and/or endovascular treatment
* Age ≥18 years

Exclusion Criteria:

* Administration of intravenous thrombolysis at another hospital in patients who are candidates for endovascular treatment
* Contraindications to intravenous thrombolysis
* Contraindications to iodinated contrast agent
* A history of ischemic stroke in three months
* Clinical diagnosis of autoimmune,inflammatory, hematological, or infectious diseases
* Clinical diagnosis of cancer
* Clinical diagnosis of severe cardiac,pulmonary,renal or liver failure
* Clinical diagnosis of dementia or psychosis
* Pregnant and lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The patients in Xijing Hospital,Yan 'an University Xianyang Hospital and Xianyang First People's Hospital
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-11-01 (Estimated); Study Completion 2023-02-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Hemorrhagic Transformation after reperfusion therapy | At 24 to 48 hours after reperfusion therapy
  Patients will undergo the cranial CT at 24 to 48 hours after reperfusion therapy to identify intracranial hemorrhage

SECONDARY OUTCOMES:
Incidence of early neurological deterioration | At 24 hours from reperfusion therapy
  Either death or an increase in the NIHSS score by ≥4 points from baseline to 24 hours after reperfusion therapy
Incidence of unfavourable short-term prognosis | At 90 days after stroke onset
  Death and major disability (modified Rankin Scale score ≥3) at 90 days after stroke onset

CONTACTS AND LOCATIONS:
Locations (1):
- Xijing Hospital, Xi'an, Shaanxi, China